CLINICAL TRIAL: NCT06187870
Title: Creation of a Bank of Biological Material From Patients and Healthy Donors (Biobank) for the Study of Urological and Uro-oncological Pathologies - URBBAN
Brief Title: Bank of Biological Material From Patients and Healthy Donors for the Study of Urological and Uro-oncological Pathologies
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Prof, IRCCS San Raffaele
Other Study IDs: URBBAN
Record Dates: First submitted 2023-12-14; First posted 2024-01-03 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Urologic Diseases; Urologic Cancer; Infertility
MeSH Terms: conditions — Urologic Diseases; Urologic Neoplasms; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of biological data — Biological samples will be collected from the patient at the time of their access to the Hospital

SUMMARY:
The project aims to collect fresh biological material derived both from surgical resections performed in diseases, neoplastic and otherwise, of urological relevance at the level of the prostate, bladder, kidney, testicle and genitourinary organs, and from peripheral blood or other fluids biological samples such as urine, seminal fluid, buccal mucosa, feces or saliva, when available.

DETAILED DESCRIPTION:
Significant studies have shown the great potential of research based on access to biobanks which has made it possible to conduct studies and obtain important results through retrospective studies carried out on samples collected some time ago. Thanks to the possibility of accessing human biological samples collected and stored in biological banks, great results have been achieved in the medical field. The project aims to collect fresh biological material deriving from surgical resections performed in neoplastic and non-neoplastic pathologies of urological relevance at the level of the prostate, bladder, kidney, testicle and genitourinary organs, both from biological samples of peripheral blood or other fluids such as urine, seminal fluid, buccal mucosa, feces or saliva, when available.

The possibility of obtaining biological samples from the patient at the time of the first visit or the first biopsy and, subsequently, in conjunction with a possible surgical intervention, could ideally give the possibility of studying the disease from its possible onset to the possible intervention, evaluating the evolution and possible association with circulating diagnostic and prognostic markers. The establishment of this collection of research material will allow access to samples of extreme value for the pathophysiological study of the disease, its origin, mechanisms and markers of progression. The data obtained can also be correlated with the patient's clinical history in order to build an overall vision potentially useful in the design of new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with an age > 18
* Ability to read and sign the informed consent
* patients affected by urological or uro-oncological diseases

Exclusion Criteria:

* People with an age < 18
* Incapacity to read and sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with urological or uro-oncological diseases and infertility
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2010-10-07 (Actual); Primary Completion 2030-10-06 (Estimated); Study Completion 2030-10-06 (Estimated)

PRIMARY OUTCOMES:
Biological sample | Baseline
  A biobank is a facility aimed at the collection, management, preservation and distribution of biomaterials and related data for research purposes

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No